CLINICAL TRIAL: NCT03642535
Title: Aminolevulinic Acid-photodynamic Therapy for Facial Actinic Keratosis Treatment and Prevention: A Long-term (3 Years) Follow-up of Prospective, Randomized, Multicenter-clinical Trial
Brief Title: Aminolevulinic Acid-photodynamic Therapy for Facial Actinic Keratosis Treatment and Prevention
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Dermatology Hospital (Other)
Collaborators: Huadong Hospital (Other); Peking University First Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); General Hospital of Ningxia Medical University (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xiuli Wang, Clinical Professor, Shanghai Dermatology Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-014
Record Dates: First submitted 2018-01-04; First posted 2018-08-22 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Actinic Keratoses
Keywords: Photodynamic Therapy; Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALA for all face group (Experimental): Scales and crusts were gently removed by curettage, and the lesions to be treated were scraped carefully to avoid bleeding. Immediately afterwards, a 1-mm thick layer of 10% ALA was applied to the all face. The area was covered with an occlusive dressing for 3 h, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's lamp. Treatment area (all face)was then separately illuminated with red light-emitting diode lamps with peak emission at 630 nm and total light dose of 100 J/cm2. The treatment is once a week for total 3 times. The patients then follow up in clinic 3 years after their treatment to have the number of actinic keratoses counted.
  Interventions: Drug: ALA
- ALA for AK lesion group (Active Comparator): Scales and crusts were gently removed by curettage, and the lesions to be treated were scraped carefully to avoid bleeding. Then a 1-mm thick layer of 10% ALA was applied to the lesion and 5 mm of surrounding healthy tissue. Vehicle control cream was applied to the non-lesion area. All area was covered with an occlusive dressing for 3 h, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's lamp. Treatment area (all face)was then separately illuminated with red light-emitting diode lamps with peak emission at 630 nm and total light dose of 100 J/cm2. The treatment is once a week for total 3 times. The patients then follow up in clinic 3 years after their treatment to have the number of actinic keratoses counted.
  Interventions: Drug: ALA

INTERVENTIONS:
Drug: ALA — In all face treatment group, a 1-mm thick layer of 10% ALA was applied to the all face; In AK lesion treatment group, a 1-mm thick layer of 10% ALA was applied to the lesion and to 5 mm of surrounding healthy tissue. And Vehicle control cream was applied to the non-lesion area.
  Other Names: Aminolevulinic Acid

SUMMARY:
Background Actinic keratoses (AKs) are often treated separately, lesion by lesion. However, in the past years, AKs have been described as a field disease and not limited to single clinically apparent lesions. Treatment should therefore target an area of field change which may treat the subclinical AKs and reduce the risk of development of further AKs, second tumours, and local recurrence.

Objectives The investigators sought to investigate whether field ALA-PDT of facial actinic keratosis would prevent new AKs, in comparison with a lesion area receiving the same ALA-PDT, in patients with clinical signs of field cancerization.

Methods Eighty patients, previously diagnosed as having AKs of the face, were randomized distribution into two groups. 10% aminolaevulinic acid (ALA)-PDT for field treatment was on one group and for a lesion area (Vehicle control cream was applied to the non-lesion area) was on the other group. During the next 5-year period of follow up, patients were clinically evaluated for new AKs.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosed with AK (OLSEN classification grade I, II, III), aged > 18 years (Because no dosing or adverse event data are currently available on the use of topical aminolevulinic acid in patients <18 years of age, children are excluded from this study);
2. All patients are unfit and reluctant to undergo surgery for any reasons, and volunteered to participate in the study and ability to understand and the willingness to sign a written informed consent. Patents are willing to pay for the treatment, and agreed to take a picture of the skin lesions.

Exclusion Criteria:

1. Those who had ALA-PDT and any other studies that affect this study within 12 weeks ;
2. There are other facial diseases that may affect the efficacy evaluation, such as other photodermatosis;
3. Take phototoxic or photosensitizer within 8 weeks;
4. Clinical and / or pathological prove that the tumor has invaded other organs or tissues;
5. Serious immunocompromised persons;
6. scar constitution;
7. Patients are known to have skin photosensitivity, porphyria, or allergies to ALA, light or lidocaine;
8. Persons are suffering from severe internal diseases, mental and mental illness, infectious diseases or pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of new Actinic Keratoses | 1, 3, 6, 9, 12, 18, 24, 30, 36 months after treatment
  The change in number of actinic keratoses at each follow-up will be measured as the primary outcome

SECONDARY OUTCOMES:
The clearance rate of Actinic Keratoses | 1 month after treatment
  The change rate in lesion clearance of Actinic Keratoses at one month after treatment will be measured as the second outcome

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Wang, PHD, MD, Study Chair — Shanghai Skin Disease Hospital
Locations (1):
- Shanghai Dermatology Hospital, Shanghai, Jingan, China

IPD SHARING:
Plan to Share IPD: Yes
underlie results
Supporting Information: CSR
Time Frame: One year after finishing this study and for permanency
Access Criteria: anyone who search pubmed
URL: http://www.ncbi.nlm.nih.gov/pubmed

REFERENCES:
- [Result] Pomerantz H, Hogan D, Eilers D, Swetter SM, Chen SC, Jacob SE, Warshaw EM, Stricklin G, Dellavalle RP, Sidhu-Malik N, Konnikov N, Werth VP, Keri J, Lew R, Weinstock MA; Veterans Affairs Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial Group. Long-term Efficacy of Topical Fluorouracil Cream, 5%, for Treating Actinic Keratosis: A Randomized Clinical Trial. JAMA Dermatol. 2015 Sep;151(9):952-60. doi: 10.1001/jamadermatol.2015.0502. PMID 25950503
- [Result] Walker JL, Siegel JA, Sachar M, Pomerantz H, Chen SC, Swetter SM, Dellavalle RP, Stricklin GP, Qureshi AA, DiGiovanna JJ, Weinstock MA. 5-Fluorouracil for Actinic Keratosis Treatment and Chemoprevention: A Randomized Controlled Trial. J Invest Dermatol. 2017 Jun;137(6):1367-1370. doi: 10.1016/j.jid.2016.12.029. No abstract available. PMID 28532759
- [Result] Perl M, Goldenberg G. Field therapy in the treatment of actinic keratosis. Cutis. 2014 Apr;93(4):172-3. No abstract available. PMID 24818175
- [Result] Stockfleth E, Gupta G, Peris K, Aractingi S, Dakovic R, Alomar A. Reduction in lesions from Lmax: a new concept for assessing efficacy of field-directed therapy for actinic keratosis. Results with imiquimod 3.75%. Eur J Dermatol. 2014 Jan-Feb;24(1):23-7. doi: 10.1684/ejd.2014.2265. PMID 24589500
- [Result] Neittaanmaki-Perttu N, Gronroos M, Tani T, Polonen I, Ranki A, Saksela O, Snellman E. Detecting field cancerization using a hyperspectral imaging system. Lasers Surg Med. 2013 Sep;45(7):410-7. doi: 10.1002/lsm.22160. PMID 24037822
- [Result] Gupta G, Stockfleth E, Peris K, Aractingi S, Alomar A, Dakovic R, Dirschka T. Long-term sustained lesion clearance from Lmax with imiquimod 3.75%, a new field-directed treatment for actinic keratosis. J Eur Acad Dermatol Venereol. 2015 Sep;29(9):1840-2. doi: 10.1111/jdv.12697. Epub 2014 Aug 29. PMID 25174261
- [Result] Pellacani G, Peris K, Guillen C, Clonier F, Larsson T, Venkata R, Puig S. A randomized trial comparing simultaneous vs. sequential field treatment of actinic keratosis with ingenol mebutate on two separate areas of the head and body. J Eur Acad Dermatol Venereol. 2015 Nov;29(11):2192-8. doi: 10.1111/jdv.13211. Epub 2015 Aug 24. PMID 26300464
- [Result] Reinhold U, Dirschka T, Ostendorf R, Aschoff R, Berking C, Philipp-Dormston WG, Hahn S, Lau K, Jager A, Schmitz B, Lubbert H, Szeimies RM. A randomized, double-blind, phase III, multicentre study to evaluate the safety and efficacy of BF-200 ALA (Ameluz((R)) ) vs. placebo in the field-directed treatment of mild-to-moderate actinic keratosis with photodynamic therapy (PDT) when using the BF-RhodoLED((R)) lamp. Br J Dermatol. 2016 Oct;175(4):696-705. doi: 10.1111/bjd.14498. Epub 2016 Jun 25. PMID 26921093
- [Result] Szeimies RM, Torezan L, Niwa A, Valente N, Unger P, Kohl E, Schreml S, Babilas P, Karrer S, Festa-Neto C. Clinical, histopathological and immunohistochemical assessment of human skin field cancerization before and after photodynamic therapy. Br J Dermatol. 2012 Jul;167(1):150-9. doi: 10.1111/j.1365-2133.2012.10887.x. Epub 2012 Jun 1. PMID 22329784
- [Result] Eibenschutz L, Silipo V, De Simone P, Buccini PL, Ferrari A, Carbone A, Catricala C. A 9-month, randomized, assessor-blinded, parallel-group study to evaluate clinical effects of film-forming medical devices containing photolyase and sun filters in the treatment of field cancerization compared with sunscreen in patients after successful photodynamic therapy for actinic keratosis. Br J Dermatol. 2016 Dec;175(6):1391-1393. doi: 10.1111/bjd.14721. Epub 2016 Oct 18. No abstract available. PMID 27167413